CLINICAL TRIAL: NCT01923675
Title: Myopia:the Role of Cone Opsin Mutations & Glasses That Control Axial Elongation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jay Neitz, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCH13693
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Myopia
Keywords: myopia; nearsightedness; axial elongation of the eye; refractive error
MeSH Terms: conditions — Myopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- color blocking tint (Experimental): Spectacles with red-blocking tint subjects will wear glasses daily for 6 months and have
  Interventions: Other: Spectacles with red-blocking tint
- holographic diffuser (Other): Spectacles with color neutral tint subjects will wear glasses daily for 6 months and have
  Interventions: Other: Spectacles with holographic diffuser and color neutral tint
- diffuser & color blocking tint (Other): Spectacles with holographic diffuser and red-blocking tint subjects will wear glasses daily for 6 months and have
  Interventions: Other: Spectacles with holographic diffuser and red-blocking tint
- holographic diffuser and neutral tint (Other): Spectacles with holographic diffuser and color neutral tint subjects will wear glasses daily for 6 months and have
  Interventions: Other: Spectacles with color neutral tint

INTERVENTIONS:
Other: Spectacles with red-blocking tint — Eyeglasses will have lenses that will correct refractive error for each subject, and will have a tint that blocks red light.
  Arms: color blocking tint
Other: Spectacles with holographic diffuser and color neutral tint — Eyeglasses will correct refractive error for each subject but will have a holographic diffuser applied to the surface and will have a color neutral filter to adjust the light intensity reaching the eyes to be the same as for groups 1 and3.
  Arms: holographic diffuser
Other: Spectacles with holographic diffuser and red-blocking tint — Eyeglasses will correct refractive error for each subject and will be tinted to block red light, and will have a holographic diffuser to blur the image.
  Arms: diffuser & color blocking tint
Other: Spectacles with color neutral tint — Eyeglasses will correct refractive error for each subject and will have a color neutral tint to adjust the light intensity reaching the eyes so it is the same as for groups 1 and 3.
  Arms: holographic diffuser and neutral tint

SUMMARY:
1. To determine the effect of spectacles with a red blocking filter on myopia progression in children.
2. To determine the effect of spectacles with a holographic diffuser that spreads incident light rays over an angle of 0.5 degrees on myopia progression in children
3. To determine the combined effects of spectacles with a red blocking filter and a diffuser that spreads incident light over an angle of 0.5 degrees on myopia progression in children.

DETAILED DESCRIPTION:
In this clinical trial we will determine whether commercially available lens tints that are normally used for cosmetic purposes or for blocking sunlight have a beneficial effect of slowing axial eye growth in children with myopia when used alone or in conjunction with a holographic diffuser that blurs the image slightly.

The following procedures will be performed on a total of 240 children from 8 to 13 years of age:

1. Color vision tests (Richmond Hardy-Rand-Rittler pseudoisochromatic plate test and/or the Rayleigh match test and/or the Neitz Test of Color Vision), and machine-based vision tests using the Titmus tester (color vision, binocularity, acuity, and heterophoria tests);
2. each subject will provide a blood sample or a buccal swab for genetic analysis of the long and middle wavelength cone photopigment genes in order to determine the relationship between the cone opsins and myopia;
3. eye measurements including axial length and corneal curvature will be performed using the Zeiss Intraocular Lens Master;
4. cycloplegic autorefraction will be doe at the beginning of the study before participants start wearing the study spectacles, after 18 months if wearing the study spectacles, and 6 months after participants stop wearing the study spectacles.

4) subjects will be randomly assigned to one of four groups, consisting of 60 subjects each, each group will be assigned one of four study spectacles.

The study spectacles for all participants will have the optimal lens corrections for both eyes.

Group 1 participants will wear spectacles with lenses tinted to blocks red light.

Group 2 participants will wear spectacles with lenses that have a holographic diffuser on surface of and that are tinted to reduce the light intensity by the same amount that the red-blocking tint does.

Group 3 participants will wear spectacles that are tinted to block red light and that have a holographic diffuser.

Group 4 participants will wear spectacles that are tinted to reduces the light intensity by the same amount that the red-blocking tint does.

Participants will wear the study glasses for 18 months. Axial length measurements will be taken twice prior to when subjects begin wearing the glasses and once every three month thereafter.

ELIGIBILITY:
Inclusion Criteria:

* nearsighted having a refractive error of at least -0.5 diopters
* myopia progression at least -.50 D per year in previous year
* astigmatism and anisometropia not more than 1.5 D
* distance monocular acuity 6/6 or better
* near monocular acuity of 0.4 M or better
* stereoacuity not more than 40 sec of arc at 40 cm
* able to respond to subjective testing
* no contact lens use during the study
* able to comply with wearing the experimental lenses daily for 18 months
* able to have axial length measurements accurately on the Zeiss Intraocular Lens Master
* willing to donate a blood sample or a buccal swab for genetic analysis
* can be refracted to 20/20 or 20/15

Exclusion Criteria:

* glaucoma, amblyopia, strabismus
* ocular disease
* developmental delay
* history of wearing bifocal lenses
* any type of eye surgery
* color vision deficiency

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-11 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Myopia progression measured by rate of axial elongation of the eye | every 3 months for 18 months
  The axial length of both eyes will be measured before wearing the experimental eyeglasses, then once every three months thereafter for 18 months, and again 6 months after subjects stop wearing the study eye glasses. The rate of axial elongation will be calculated.

SECONDARY OUTCOMES:
Myopia progression measured by cycloplegic autorefraction. | 18 months
  A cycloplegic autorefraction will be done at the beginning of the study before subjects start wearing the study glasses, after 18 months of wearing the study glasses,and again about 6 months after wearing the study glasses stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Neitz, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Carkeet A, Saw SM, Gazzard G, Tang W, Tan DT. Repeatability of IOLMaster biometry in children. Optom Vis Sci. 2004 Nov;81(11):829-34. doi: 10.1097/01.opx.0000145020.33250.c0. PMID 15545808
- [Background] Congdon NG, Friedman DS, Lietman T. Important causes of visual impairment in the world today. JAMA. 2003 Oct 15;290(15):2057-60. doi: 10.1001/jama.290.15.2057. No abstract available. PMID 14559961
- [Background] Grosvenor T. Why is there an epidemic of myopia? Clin Exp Optom. 2003 Sep;86(5):273-5. doi: 10.1111/j.1444-0938.2003.tb03122.x. No abstract available. PMID 14558848
- [Background] Gwiazda J, Hyman L, Hussein M, Everett D, Norton TT, Kurtz D, Leske MC, Manny R, Marsh-Tootle W, Scheiman M. A randomized clinical trial of progressive addition lenses versus single vision lenses on the progression of myopia in children. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1492-500. doi: 10.1167/iovs.02-0816. PMID 12657584
- [Background] Ip JM, Rose KA, Morgan IG, Burlutsky G, Mitchell P. Myopia and the urban environment: findings in a sample of 12-year-old Australian school children. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):3858-63. doi: 10.1167/iovs.07-1451. Epub 2008 May 9. PMID 18469186
- [Background] Rein DB, Zhang P, Wirth KE, Lee PP, Hoerger TJ, McCall N, Klein R, Tielsch JM, Vijan S, Saaddine J. The economic burden of major adult visual disorders in the United States. Arch Ophthalmol. 2006 Dec;124(12):1754-60. doi: 10.1001/archopht.124.12.1754. PMID 17159036
- [Background] Saw SM, Gazzard G, Shih-Yen EC, Chua WH. Myopia and associated pathological complications. Ophthalmic Physiol Opt. 2005 Sep;25(5):381-91. doi: 10.1111/j.1475-1313.2005.00298.x. PMID 16101943
- [Background] Saw SM, Katz J, Schein OD, Chew SJ, Chan TK. Epidemiology of myopia. Epidemiol Rev. 1996;18(2):175-87. doi: 10.1093/oxfordjournals.epirev.a017924. No abstract available. PMID 9021311
- [Background] Vitale S, Sperduto RD, Ferris FL 3rd. Increased prevalence of myopia in the United States between 1971-1972 and 1999-2004. Arch Ophthalmol. 2009 Dec;127(12):1632-9. doi: 10.1001/archophthalmol.2009.303. PMID 20008719